CLINICAL TRIAL: NCT05543174
Title: An Open-Label, Phase 3 Study to Evaluate the Efficacy and Safety of TAK-625 in the Treatment of Subjects With Alagille Syndrome
Brief Title: A Study of TAK-625 for the Treatment of Alagille Syndrome (ALGS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-625-3001; jRCT2051220098 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Alagille Syndrome (ALGS)
MeSH Terms: conditions — Alagille Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TAK-625 (Experimental): TAK-625 200 mcg per kilogram, orally, once daily for 1 week. After that, TAK-625 400 mcg per kilogram, orally, once daily after Week 1.
  Interventions: Drug: TAK-625

INTERVENTIONS:
Drug: TAK-625 — TAK-625 200 mcg or 400 mcg per kilogram, orally, once daily
  Other Names: Maralixibat chloride

SUMMARY:
The main aim of the study is to check if TAK-625 improves symptoms of Alagille Syndrome (ALGS), side effect from the study treatment or TAK-625, and how much TAK-625 stays in their blood over time. This will help the study sponsor (Takeda) to work out the best dose to give people in the future.

The participants will be treated with TAK-625 for up to the end of study (about 34 months).

Participants will visit their study clinic 9 times from the start of study. After 9 times visits, participants will visit their study clinic every 12 weeks up to the end of study.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is Japanese male or female with a body weight >=3.0 kilograms (kg) and who is >=1 month of age at the time of informed consent.
2. The participant is diagnosed with ALGS.
3. The participant has one or more of the following evidences of cholestasis:

   1. Total serum bile acid (sBA) >3^ upper limit of the normal range (ULN) for age.
   2. Direct bilirubin (conjugated) >1 mg/dL.
   3. Lipid soluble vitamin (LSV) deficiency otherwise unexplainable.
   4. Gamma-glutamyl transferase (GGT) >3^ ULN for age.
   5. Intractable pruritus explainable only by liver disease.
4. The participant is expected to have a consistent caregiver(s) for the duration of the study.
5. The participant has an access to phone for scheduled calls from study site.
6. Both a caregiver and participant above the age of assent are capable of reading and understanding the questionnaires.
7. Caregivers (and age-appropriate participants) must be willing and able to use an eDiary device during the study.
8. Caregivers (and age-appropriate participants) must complete at least 10 eDiary reports (morning or evening) during each of 2 consecutive weeks of the screening period (maximum possible reports=14 per week), even if the participant is an adult (over 18 years old).
9. Average daily score >2 on the ItchRO questionnaire (maximum possible daily score of 4) for 2 consecutive weeks in the screening period, prior to dosing. A daily score is the higher of the scores for the morning and evening ItchRO. The average daily score is the sum of all daily scores divided by the number of days the ItchRO was completed. Since it is difficult to evaluate pruritus in infants, participants <12 months of age at screening whose pruritus is unavoidably difficult to be evaluated are not necessarily required to meet the above score.

Exclusion Criteria:

1. The participant has chronic diarrhea requiring ongoing intravenous (IV) fluid or nutritional intervention.
2. The participant has a previous history of surgical interruption of the enterohepatic circulation.
3. The participant has a previous liver transplant.
4. The participant decompensated cirrhosis (ALT >15^ ULN, international normalized ratio [INR] >1.5 [unresponsive to vitamin K therapy], albumin <3.0 g/dL, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy).
5. The participant has a history or presence of other concomitant liver disease.
6. The participant has a history or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, including bile salt metabolism in the intestine (eg, inflammatory bowel disease).
7. The participant has a history or presence of gallstones or kidney stones.
8. The participant has a possible malignant liver mass in imaging, including screening ultrasound.
9. The participant has cancers, except for in situ carcinoma, or cancers treated at least 5 years prior to screening with no evidence of recurrence.
10. The participant has received bile acid/lipid binding resins or IBAT inhibitors within 28 days prior to screening and throughout the trial.
11. The participant who has received sodium phenylbutyrate for less than 6 months at the initiation of screening.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2025-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Japan (8):
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Miyagi Children's Hospital, Sendai, Miyagi
  - Kindai University Nara Hospital, Ikoma, Nara
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Kyoto University Hospital, Kyoto
  - Saitama Prefectural Children's Medical Center, Saitama

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/183b4344d3af4327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 sites in Japan.
Pre-assignment Details: Participants diagnosed with Alagille Syndrome (ALGS) were enrolled to receive TAK-625 once daily (QD). The study consisted of the screening period, 2-week dose escalation period, 46-week stable dosing period, a follow-up dosing period after Week 48, and a safety follow-up period.
Groups:
- TAK-625: Participants diagnosed with ALGS received TAK-625 orally, QD. In dose escalation period, dose was increased weekly, 200 micrograms per kilograms (mcg/kg) and 400 mcg/kg for up to 2 weeks. After the dose escalation period, each participant continued dosing with TAK-625 400 mcg/kg, orally, QD dose level in the stable dosing period for 46 weeks and a follow-up dosing period after Week 48, followed by a safety follow-up period.
Period: Overall Study
Arm/Group | TAK-625
Started | 7
Dosed TAK-625 200 mcg/kg (TAK-625 orally, QD for 1 week in Dose Escalation Period.) | 7
Dosed TAK-625 400 mcg/kg (TAK-625 orally, QD for 1 week in Dose Escalation Period and for up to 46 weeks in the stable dosing period and a follow-up dosing period after Week 48, followed by a safety follow-up period.) | 7
Completed | 6
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) included all participants who received at least one dose of study drug. As per-planned analysis, the data for baseline measures were collected, analyzed and reported as a single cohort.
Groups:
- TAK-625: Participants diagnosed with ALGS received TAK-625 orally, QD. In dose escalation period, dose was increased weekly, 200 mcg/kg and 400 mcg/kg for up to 2 weeks. After the dose escalation period, each participant continued dosing with TAK-625 400 mcg/kg, orally, QD dose level in the stable dosing period for 46 weeks and a follow-up dosing period after Week 48, followed by a safety follow-up period.
Arm/Group | TAK-625
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.143 (3.8675)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Fasting Serum Bile Acid (sBA) Levels From Week 18 to Week 22
Description: Change in fasting sBA levels from Week 18 to 22 was reported. Change was calculated as: observed value at Week 22- observed value at Week 18.
Time Frame: From Week 18 to Week 22
Population: ITT included all participants who received at least one dose of study drug. As per-planned analysis, the data for outcome measure were collected, analyzed and reported as a single cohort.
Measure: Mean (95% Confidence Interval); unit: micromoles per liter (mcmol/L)
Arm/Group | TAK-625
Number analyzed (Participants) | 7
micromoles per liter (mcmol/L) | 17.643 [-31.6389 to 66.9246]

2. Secondary Outcome: Change in Fasting sBA Levels From Baseline to Week 18
Description: Change in fasting sBA levels from baseline to Week 18 was reported. Change was calculated as: observed value at Week 18 - observed value at baseline (before dosing).
Time Frame: Baseline to Week 18
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mcmol/L
Arm/Group | TAK-625
Number analyzed (Participants) | 7
mcmol/L | 8.300 [-37.4110 to 54.0110]

3. Secondary Outcome: Change in Weekly Average Severity of Pruritus Measured by Itch Reported Outcome (ItchRO) (Observer Instrument [Obs]) From Baseline to Week 18
Description: The ItchRO (Obs) scale measures severity of pruritus. The score on ItchRO (Obs) scale ranged from 0 to 4, where 0=None observed or reported, 1=Mild, 2=Moderate, 3=Severe, 4=Very severe. A higher score indicated more severe pruritus. Weekly average severity of Pruritus is calculated based on daily maximum of morning and evening severity scores measured by ItchRO (Obs). Weekly average severity was calculated as the average of the daily maximum of morning and evening over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 18 (Day 120 to Day 126) - average value of baseline (Day -7 to Day -1).
Time Frame: Baseline to Week 18
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 7
score on a scale | -1.531 [-2.3405 to -0.7208]

4. Secondary Outcome: Change in Weekly Average Morning Severity of Pruritus Measured by Itch Reported Outcome (ItchRO) (Observer Instrument [Obs]) From Baseline to Week 18
Description: The ItchRO (Obs) scale measures severity of pruritus. The score on ItchRO (Obs) scale ranged from 0 to 4, where 0=None observed or reported, 1=Mild, 2=Moderate, 3=Severe, 4=Very severe. A higher score indicated more severe pruritus. Weekly average morning severity was calculated as the average of the daily morning scores over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 18 (Day 120 to Day 126) - average value of baseline (Day -7 to Day -1).
Time Frame: Baseline to Week 18
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 7
score on a scale | -1.327 [-2.1071 to -0.5460]

5. Secondary Outcome: Change in Weekly Average Severity of Pruritus Measured by ItchRO (Obs) From Week 18 to Week 22
Description: The ItchRO (Obs) scale measures severity of pruritus. The score on ItchRO (Obs) scale ranged from 0 to 4, where 0=None observed or reported, 1=Mild, 2=Moderate, 3=Severe, 4=Very severe. A higher score indicated more severe pruritus. Weekly average severity of Pruritus was calculated based on daily maximum of morning and evening severity scores measured by ItchRO (Obs). Weekly average severity were calculated as the average of the daily maximum of morning and evening over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 22 (Day 148 to Day 154) - average value of Week 18 (Day 120 to Day 126).
Time Frame: From Week 18 to Week 22
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 7
score on a scale | -0.286 [-0.6594 to 0.0880]

6. Secondary Outcome: Change in Weekly Average Morning Severity of Pruritus Measured by ItchRO (Obs) From Week 18 to Week 22
Description: The ItchRO (Obs) scale measures severity of pruritus. The score on ItchRO (Obs) scale ranged from 0 to 4, where 0=None observed or reported, 1=Mild, 2=Moderate, 3=Severe, 4=Very severe. A higher score indicated more severe pruritus. Weekly average morning severity was calculated as the average of the daily morning scores over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 22 (Day 148 to Day 154) - average value of Week 18 (Day 120 to Day 126).
Time Frame: From Week 18 to Week 22
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 7
score on a scale | -0.280 [-0.6769 to 0.1163]

7. Secondary Outcome: Change in Weekly Average Severity of Pruritus Measured by ItchRO (Pt) From Baseline to Week 18
Description: The ItchRO (Pt) scale measures severity of pruritus. The score on ItchRO (Pt) scale ranged from 0 to 4, where 0= Not felt itchy, 1= Felt a little bit itchy, 2= Felt pretty itchy, 3= Felt very itchy, 4= Felt very, very itchy. A higher score indicated more severe pruritus. Weekly average severity of Pruritus was calculated based on daily maximum of morning and evening severity scores measured by ItchRO (Pt). Weekly average scores was calculated as the average of the daily maximum of morning and evening over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 18 (Day 120 to Day 126) - average value of baseline (Day -7 to Day -1).
Time Frame: Baseline to Week 18
Population: ITT included all participants who received at least one dose of study drug. As per-planned analysis, the data for outcome measure were collected, analyzed and reported as a single cohort. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 3
score on a scale | -1.381 [-5.0058 to 2.2439]

8. Secondary Outcome: Change in Weekly Average Morning Severity of Pruritus Measured by ItchRO (Pt) From Baseline to Week 18
Description: The ItchRO (Pt) scale measures severity of pruritus. The score on ItchRO (Pt) scale ranged from 0 to 4, where 0= Not felt itchy, 1= Felt a little bit itchy, 2= Felt pretty itchy, 3= Felt very itchy, 4= Felt very, very itchy. A higher score indicated more severe pruritus. Weekly average morning severity was calculated as the average of the daily morning scores over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 18 (Day 120 to Day 126) - average value of baseline (Day -7 to Day -1).
Time Frame: Baseline to Week 18
Population: ITT included all participants who received at least one dose of study drug. Here, "overall number of participants analyzed" signified those participants who were evaluable for this outcome measure. As per-planned analysis, the data for outcome measure were collected, analyzed and reported as a single cohort.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 3
score on a scale | -1.238 [-3.6537 to 1.1775]

9. Secondary Outcome: Change in Alanine Aminotransferase (ALT) and Alkaline Phosphatase (ALP) Levels From Baseline to Week 18
Description: Change in ALT and ALP levels from baseline to Week 18 were reported. Change was calculated as: observed value at Week 18 - observed value at baseline (before dosing).
Time Frame: Baseline to Week 18
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Units per liter (U/L)
Arm/Group | TAK-625
Number analyzed (Participants) | 7
Units per liter (U/L)
  Change in ALT | 17.7 [-52.66 to 88.09]
  Change in ALP | 75.6 [-186.50 to 337.64]

10. Secondary Outcome: Change in Bilirubin (Total and Direct) Levels From Baseline to Week 18
Description: Change in bilirubin (total and direct) from baseline to Week 18 was reported. Change was calculated as: observed value at Week 18 - observed value at baseline (before dosing).
Time Frame: Baseline to Week 18
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mcmol/L
Arm/Group | TAK-625
Number analyzed (Participants) | 7
mcmol/L
  Change in total bilirubin | 11.3619 [-20.13472 to 42.85861]
  Change in direct bilirubin | 8.6009 [-15.59872 to 32.80046]

11. Secondary Outcome: Change in Weekly Average Severity of Pruritus Measured by ItchRO (Pt) From Week 18 to Week 22
Description: The ItchRO (Pt) scale measures severity of pruritus. The score on ItchRO (Pt) scale ranged from 0 to 4, where 0= Not felt itchy, 1= Felt a little bit itchy, 2= Felt pretty itchy, 3= Felt very itchy, 4= Felt very, very itchy. A higher score indicated more severe pruritus. Weekly average severity of Pruritus was calculated based on daily maximum of morning and evening severity scores measured by ItchRO (Pt). Weekly average scores was calculated as the average of the daily maximum of morning and evening over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 22 (Day 148 to Day 154) - average value of Week 18 (Day 120 to Day 126).
Time Frame: From Week 18 to 22
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 3
score on a scale | 0.000 [-0.6147 to 0.6147]

12. Secondary Outcome: Change in Weekly Average Morning Severity of Pruritus Measured by ItchRO (Pt) From Week 18 to Week 22
Description: The ItchRO (Pt) scale measures severity of pruritus. The score on ItchRO (Pt) scale ranged from 0 to 4, where 0= Not felt itchy, 1= Felt a little bit itchy, 2= Felt pretty itchy, 3= Felt very itchy, 4= Felt very, very itchy. A higher score indicated more severe pruritus. Weekly average morning severity was calculated as the average of the daily morning scores over the visit consisting of the 7 days on or before the scheduled Study Day (i.e., the sum of the scores divided by the number of non-missing scores). Change was calculated as: average value of Week 22 (Day 148 to Day 154) - average value of Week 18 (Day 120 to Day 126).
Time Frame: From Week 18 to 22
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TAK-625
Number analyzed (Participants) | 3
score on a scale | -0.032 [-0.4120 to 0.3485]

13. Secondary Outcome: Change in ALT and ALP Levels From Week 18 to 22
Description: Change in ALT and ALP from Week 18 to 22 was reported. Change was calculated as: observed value at Week 22 - observed value at Week 18.
Time Frame: From Week 18 to 22
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | TAK-625
Number analyzed (Participants) | 7
U/L
  Change in ALT | 7.9 [-22.18 to 37.89]
  Change in ALP | -32.3 [-79.12 to 14.55]

14. Secondary Outcome: Change in Bilirubin (Total and Direct) Levels From Week 18 to 22
Description: Change in bilirubin (total and direct) from Week 18 to 22 was reported. Change was calculated as: observed value at Week 22 - observed value at Week 18.
Time Frame: From Week 18 to 22
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mcmol/L
Arm/Group | TAK-625
Number analyzed (Participants) | 7
mcmol/L
  Change in total bilirubin | 0.6842 [-4.60580 to 5.97412]
  Change in direct bilirubin | 1.2217 [-1.83803 to 4.28146]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to Week 133
Description: As per-planned analysis, the data for adverse events section were collected, analyzed and reported as a single cohort.
Arm/Group | TAK-625
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-625 (N=7)
Liver transplant (Surgical and medical procedures) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Weight gain poor (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-625 (N=7)
Administration site extravasation (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Anal rash (Gastrointestinal disorders) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
COVID-19 (Infections and infestations) | 1
Chapped lips (Gastrointestinal disorders) | 1
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1
Defaecation urgency (Gastrointestinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eyelid injury (Injury, poisoning and procedural complications) | 1
Gastroenteritis (Infections and infestations) | 1
Hand-foot-and-mouth disease (Infections and infestations) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 1
Ocular hyperaemia (Eye disorders) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rhinitis (Infections and infestations) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT05543174/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT05543174/SAP_002.pdf